CLINICAL TRIAL: NCT00018876
Title: Radiotherapy to Prevent Fibrosis After Lumbar Laminectomy
Brief Title: Low-Dose Radiation to Prevent Complications of Back Surgery
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: R21AR047121 (NIH); R21AR047121 (NIH); NIAMS-057
Record Dates: First submitted 2001-07-05; First posted 2001-07-09 (Estimated); Last update posted 2013-06-07 (Estimated); Status verified 2006-03

CONDITIONS: Failed Back Surgery Syndrome; Postlaminectomy Syndrome; Postdiscectomy Epidural Fibrosis
Keywords: Epidural fibrosis; Failed back surgery syndrome; Postlaminectomy syndrome; Lumbar laminectomy; Radiotherapy; Radiation; Perineural scar formation; Peridural fibrosis; Back surgery
MeSH Terms: conditions — Failed Back Surgery Syndrome; post laminectomy syndrome

INTERVENTIONS:
Procedure: Lumbar nerve root decompression
Procedure: Preoperative low-dose external beam radiation

SUMMARY:
More than 10,000 people each year in the United States have "failed back surgery syndrome" caused by scars that form around the outer surface of the spinal cord. Such scarring, known as peridural fibrosis, is common after back surgery known as either lumbar discectomy or laminectomy. Peridural fibrosis may cause recurring low back pain or leg pain after surgery. Operating again to remove the scar tissue often leads to more scarring.

Researchers have not previously studied radiation as a way to prevent peridural fibrosis. We will test whether low-dose radiation given 24 hours before surgery will decrease the amount of peridural fibrosis and if this reduction will lead to improved results of surgery. Half of the participants will receive radiation before surgery and the other half will not. We will evaluate patients at followup visits 1, 3, 6, and 12 months after surgery with a physical exam and questionnaire. At 12 months, we will obtain magnetic resonance imaging (MRI) of the lower spine.

DETAILED DESCRIPTION:
Researchers have long known that low-dose radiation inhibits fibroblast and osteoblast activity. Studies in humans have shown that perioperative radiation therapy is a useful way to prevent both keloid and heterotopic bone formation. However, researchers have not previously studied radiation as a means to inhibit peridural fibrosis. Our previous studies of both rat and dog models showed a significant reduction in peridural fibrosis after laminectomy using low-dose external beam radiation (700 cGy) given 24 hours prior to surgery. Based on our results from these animal studies, we will test whether (1) low-dose radiation given 24 hours before surgery will decrease the amount of peridural fibrosis in people and (2) this reduction in peridural fibrosis will lead to improved results of surgery.

For this study, we will enroll 46 patients with failed back surgery syndrome believed to be secondary to perineural fibrosis in a randomized, double-blinded, controlled clinical trial. We will assign patients to one of two groups before surgery: preoperative radiation (treatment group) or no preoperative radiation (control group). We will treat half of the patients with external beam radiation before re-exploration and decompression of their peridural fibrosis (treatment group) and perform re-exploration and decompression in the other half without preoperative radiation (control group).

All patients will undergo simulation radiation treatment planning and will not know if they received radiation or not. For patients randomized to receive preoperative radiation, we will administer a single dose of 700 cGy to a 6.0-cm-wide field centered on the spinal cord at the affected level, using a 6 MV Varian 600C linear accelerator. We will administer treatment with two fields angled 45 degrees from the vertical plane so that the skin surface for the proposed incision will not be irritated. This should prevent any wound healing problems. Only the radiation oncologist and research assistant will know whether radiation was administered. The patient and the surgeon will be masked as to the treatment.

The neurosurgeon co-investigators will perform the same surgical procedure on all patients 24 hours after their radiation (or sham) treatment. We will give all patients preoperative antibiotics. The surgeon will reopen the previous midline posterior lumbar skin incision and dissect the subcutaneous tissue away from the spinous process and laminae. Once the surgeon has adequately exposed the previous surgical site, he or she will place a self-retaining retractor. The surgeon will decompress the nerve by removing the scar tissue from around the nerve root and thecal sac. The surgeon will also remove any intravertebral disc material thought to be causing nerve root compression. On completion of the operation, the surgeon will stop bleeding with electrocautery, irrigate the wound with antibiotic, and close the wound in layers. In general, the hospital stay after surgery is one night. The patient begins gradual ambulation on the evening of surgery.

We will administer the North American Spine Society (NASS) Lumbar Spine Outcome Assessment to patients before treatment and at followup visits to assess their physical functioning. We will also use the NASS questionnaire to collect demographic and lifestyle information at baseline and to assess patient expectations regarding treatment and level of satisfaction with the treatment during the followup period. We will do a physical examination and administer the patient-reported questionnaire prior to surgery and at 1, 3, 6, and 12 months after surgery. We will obtain magnetic resonance (MR) imaging of the lumbar spine 12 months after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a clinical diagnosis of failed back surgery syndrome.
* Previous surgery at either the L4-5 or L5-S1 levels.
* Patients with peridural fibrosis around the symptomatic nerve root (either L5 or S1) on contrast-enhanced MR imaging.
* Willing and able to be treated and followed at the University of Pittsburgh Medical Center.
* Cooperative individuals with no language barrier, and who sign an informed consent form.

Exclusion Criteria:

* Patients less than 18 years of age.
* Patients with prior radiotherapy to the same region of the back.
* Female patients with a functioning, intact reproductive system are ineligible until a pregnancy test performed within 48 hours of radiotherapy rules out pregnancy.
* Patients with organic brain syndrome or dementia.
* Severe vascular, pulmonary or coronary artery disease which would place them at an unacceptably high risk to undergo general anesthesia.
* Myocardial infarction within the last 6 months.
* Metastatic cancer.
* Excessive alcohol consumption or evidence of drug use.
* Spondylolisthesis requiring surgical fusion (greater than 5 mm of vertebral slippage.)
* Unable to undergo MR imaging.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46
Dates: Start 2000-10; Study Completion 2002-10

CONTACTS AND LOCATIONS:
Overall Officials: Peter C. Gerszten, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Background] Abitbol JJ, Lincoln TL, Lind BI, Amiel D, Akeson WH, Garfin SR. Preventing postlaminectomy adhesion. A new experimental model. Spine (Phila Pa 1976). 1994 Aug 15;19(16):1809-14. doi: 10.1097/00007632-199408150-00004. PMID 7973979
- [Background] Brotchi J, Pirotte B, De Witte O, Levivier M. Prevention of epidural fibrosis in a prospective series of 100 primary lumbo-sacral discectomy patients: follow-up and assessment at re-operation. Neurol Res. 1999;21 Suppl 1:S47-50. doi: 10.1080/01616412.1999.11741027. PMID 10214572
- [Background] Daltroy LH, Cats-Baril WL, Katz JN, Fossel AH, Liang MH. The North American spine society lumbar spine outcome assessment Instrument: reliability and validity tests. Spine (Phila Pa 1976). 1996 Mar 15;21(6):741-9. doi: 10.1097/00007632-199603150-00017. PMID 8882698
- [Background] Dullerud R, Graver V, Haakonsen M, Haaland AK, Loeb M, Magnaes B. Influence of fibrinolytic factors on scar formation after lumbar discectomy. A magnetic resonance imaging follow-up study with clinical correlation performed 7 years after surgery. Spine (Phila Pa 1976). 1998 Jul 1;23(13):1464-9. doi: 10.1097/00007632-199807010-00007. PMID 9670398
- [Background] Fandino J, Botana C, Viladrich A, Gomez-Bueno J. Reoperation after lumbar disc surgery: results in 130 cases. Acta Neurochir (Wien). 1993;122(1-2):102-4. doi: 10.1007/BF01446994. PMID 8333299
- [Background] Geisler FH. Prevention of peridural fibrosis: current methodologies. Neurol Res. 1999;21 Suppl 1:S9-22. doi: 10.1080/01616412.1999.11741021. PMID 10214566
- [Background] Gerszten PC, Moossy JJ, Bahri S, Kalend A, Martinez AJ. Inhibition of peridural fibrosis after laminectomy using low-dose external beam radiation in a rat model. Neurosurgery. 1999 Mar;44(3):597-602; discussion 602-3. doi: 10.1097/00006123-199903000-00090. PMID 10069597
- [Background] Grane P, Tullberg T, Rydberg J, Lindgren L. Postoperative lumbar MR imaging with contrast enhancement. Comparison between symptomatic and asymptomatic patients. Acta Radiol. 1996 May;37(3 Pt 1):366-72. doi: 10.1177/02841851960371P177. PMID 8845271
- [Background] Hinton JL Jr, Warejcka DJ, Mei Y, McLendon RE, Laurencin C, Lucas PA, Robinson JS Jr. Inhibition of epidural scar formation after lumbar laminectomy in the rat. Spine (Phila Pa 1976). 1995 Mar 1;20(5):564-70; discussion 579-80. doi: 10.1097/00007632-199503010-00011. PMID 7604326
- [Background] Jonsson B, Stromqvist B. Repeat decompression of lumbar nerve roots. A prospective two-year evaluation. J Bone Joint Surg Br. 1993 Nov;75(6):894-7. doi: 10.1302/0301-620X.75B6.8245078.
- [Background] Lo TC, Seckel BR, Salzman FA, Wright KA. Single-dose electron beam irradiation in treatment and prevention of keloids and hypertrophic scars. Radiother Oncol. 1990 Nov;19(3):267-72. doi: 10.1016/0167-8140(90)90153-n. PMID 2126387
- [Background] Long DM. Failed back surgery syndrome. Neurosurg Clin N Am. 1991 Oct;2(4):899-919. PMID 1840393
- [Background] Maroon JC, Abla A, Bost J. Association between peridural scar and persistent low back pain after lumbar discectomy. Neurol Res. 1999;21 Suppl 1:S43-6. doi: 10.1080/01616412.1999.11741026. PMID 10214571
- [Background] Nguyen CM, Haughton VM, Ho KC, An HS. MR contrast enhancement: an experimental study in postlaminectomy epidural fibrosis. AJNR Am J Neuroradiol. 1993 Jul-Aug;14(4):997-1002. PMID 8352176
- [Background] North RB, Campbell JN, James CS, Conover-Walker MK, Wang H, Piantadosi S, Rybock JD, Long DM. Failed back surgery syndrome: 5-year follow-up in 102 patients undergoing repeated operation. Neurosurgery. 1991 May;28(5):685-90; discussion 690-1. PMID 1831546
- [Background] Porchet F, Lombardi D, de Preux J, Pople IK. Inhibition of epidural fibrosis with ADCON-L: effect on clinical outcome one year following re-operation for recurrent lumbar radiculopathy. Neurol Res. 1999;21 Suppl 1:S51-60. doi: 10.1080/01616412.1999.11741028. PMID 10214573
- [Background] Ross JS, Robertson JT, Frederickson RC, Petrie JL, Obuchowski N, Modic MT, deTribolet N. Association between peridural scar and recurrent radicular pain after lumbar discectomy: magnetic resonance evaluation. ADCON-L European Study Group. Neurosurgery. 1996 Apr;38(4):855-61; discussion 861-3. PMID 8692415
- [Background] Yukawa Y, Kato F, Kajino G, Nakamura S. Serial gadolinium-enhanced MR imaging after lumbar disc resection: observation of the affected root. J Spinal Disord. 1997 Oct;10(5):404-9. PMID 9355057
- [Result] Gerszten PC, Moossy JJ, Flickinger JC, Welch WC. Low-dose radiotherapy for the inhibition of peridural fibrosis after reexploratory nerve root decompression for postlaminectomy syndrome. J Neurosurg. 2003 Oct;99(3 Suppl):271-7. doi: 10.3171/spi.2003.99.3.0271. PMID 14563144